CLINICAL TRIAL: NCT02465541
Title: Lifestyle Interventions to Improve Physical Function and Quality of Life in Endometrial Cancer Survivors: The Role of a Gentle Yoga Based Exercise Program
Brief Title: Gentle Yoga and Dietary Counseling in Improving Physical Function and Quality of Life in Stage I-II Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brian Focht, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-13005; NCI-2014-00770 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-05-16; First posted 2015-06-08 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Endometrial Carcinoma
Keywords: Cancer Survivors; Yoga; Endometrial Cancer
MeSH Terms: conditions — Obesity; Endometrial Neoplasms | interventions — Yoga; Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (gentle yoga and dietary counseling) (Experimental): Participants undergo onsite gentle yoga once weekly over 45-60 minutes for 8 weeks and home-based gentle yoga for 6 weeks. Participants also undergo dietary counseling over 8 weeks.
  Interventions: Procedure: Gentle yoga therapy; Other: counseling intervention; Other: quality-of-life assessment; Other: questionnaire administration
- Arm II (enhanced usual care) (Active Comparator): Participants undergo enhanced usual care designed to educate on best practices for exercise, diet and lifestyle change once weekly for 14 weeks.
  Interventions: Other: educational intervention; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Procedure: Gentle yoga therapy — Mindfulness in Motion is a mindfulness based intervention that is an 8-10 week program for adults interested in learning a practical strategy for stress reduction, intended to be delivered on the worksite or home.
  Other Names: yoga
  Arms: Arm I (gentle yoga and dietary counseling)
Other: counseling intervention — Undergo dietary counseling that will include 10 (20-min) nutritional counseling sessions with a registered dietitian.
  Other Names: counseling and communications studies
  Arms: Arm I (gentle yoga and dietary counseling)
Other: educational intervention — Undergo enhanced usual care
  Other Names: intervention, educational
  Arms: Arm II (enhanced usual care)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well gentle yoga and dietary counseling lifestyle change effects physical function and quality of life of endometrial cancer survivors. Gentle yoga and dietary counseling may help improve physical function and quality of life for stage I-II endometrial cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and efficacy of a combined lifestyle intervention (yoga + diet) to positively impact physical function and quality of life for endometrial cancer survivors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Participants undergo onsite gentle yoga once weekly over 45-60 minutes for 8 weeks and home-based gentle yoga for 6 weeks. Participants also undergo dietary counseling over 8 weeks.

ARM II: Participants undergo enhanced usual care designed to educate on best practices for exercise, diet and lifestyle change once weekly for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Previous diagnosis of grade 1 or 2, stage I or II endometrioid endometrial cancers ("type I cancers") as confirmed during surgical intervention for treatment
* Overweight or obese (> 25 kg/m^2)
* Anytime from treatment
* Treating oncologist consent
* Primary physician consent to engage in physical activity unsupervised
* Ambulatory or able to engage in walking for at least 15 minutes
* Sedentary lifestyle, as engaging in less than 100 minutes structured aerobic walking, cycling or swimming per week

Exclusion Criteria:

* No prior type I endometrial cancer diagnosis
* Prior diagnosis of other cancer
* Currently (previous 6 months) engaged in structured exercise either aerobic or yoga based
* Severe heart or systemic disease: evidence of documented myocardial infarction, chronic unstable angina, symptomatic congestive heart failure, uncontrolled hypertension
* Severe musculoskeletal disease: severe muscle or joint disorders due to disease or trauma, amputations, or any condition that significantly impair physical capabilities, as defined by the physician
* Non-ambulatory
* Concurrent diagnosis of organic brain syndrome, dementia, mental retardation, or significant sensory deficit
* Major mental illness (e.g., schizophrenia, major depressive disorder)
* Unwilling to give consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Examine change from baseline in physical function as measured by the Short Physical Performance Battery (SPPB). | Up to 14 weeks
  Physical function will be assess using a SPPB walk performance assessment. Quality life will be assessed via the SF-36 and the Functional Assessment of Cancer Therapy-Endometrial FACT-EN.

SECONDARY OUTCOMES:
Examine intervention feasibility using a composite assessment. | Up to 14 weeks
  Descriptive statistics for the feasibility measures will be calculated using recruitment, adherence, and retention rate.

OTHER OUTCOMES:
Change from baseline in quality of life as measured by the FACT-G (Functional Assessment of Cancer Therapy: General) | Up to 14 weeks
Change from baseline in mindfulness as measured by the 5 Factor mindfulness questionnaires (FFMQ) | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Focht, PhD, FACSM, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu